CLINICAL TRIAL: NCT05505409
Title: Efficacy, Safety, Immune Function of Pirfenidone in the Treatment of Connetive Tissue Disease -Related Interstitial Lung Disease(CTD-LID)
Brief Title: Efficacy and Safety of Pirfenidone in CTD-ILD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Qiang Shu, Principal Investigator, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PFD-CTD-ILD QiluH
Record Dates: First submitted 2022-08-16; First posted 2022-08-17 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Pirfenidone; Connective Tissue Diseases; Interstitial Lung Disease
Keywords: pirfenidone; interstitial lung disease; connective tissue disease; rheumatoid arthritis; systemic sclerosis; inflammatory myopathy
MeSH Terms: conditions — Connective Tissue Diseases; Lung Diseases, Interstitial; Arthritis, Rheumatoid; Scleroderma, Systemic; Myositis | interventions — pirfenidone; Glucocorticoids; Immunosuppressive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pirfenidone group (Experimental): CTD-ILD patients treated with pirfenidone、glucocorticoid and immunosuppressant.
  Interventions: Drug: Pirfenidone; Drug: glucocorticoid and immunosuppressant
- No-pirfenidone group (Active Comparator): CTD-ILD patients treated with glucocorticoid and immunosuppressant,without pirfebidone
  Interventions: Drug: glucocorticoid and immunosuppressant

INTERVENTIONS:
Drug: Pirfenidone — Drug:pirfenidone CTD-ILD patients treated with pirfenidone up to the maximum tolerable dose Drug: glucocorticoid and immunosuppressant CTD-ILD patients treated with glucocorticoid and immunosuppressant according to the condition of the disease
  Other Names: glucocorticoid and immunosuppressant
  Arms: pirfenidone group
Drug: glucocorticoid and immunosuppressant — Drug: glucocorticoid and immunosuppressant CTD-ILD patients treated with glucocorticoid and immunosuppressant according to the condition of the disease

SUMMARY:
A single-center randomized controlled study will be used to observe the efficacy and safety of pirfenidone on CTD-ILD patients for 24 months.

The main research endpoints is the lung function (FVC) at 6 months. The clinical dyspnea score, 6-minute walking distance, index of lung function and imaging indicators are evaluated, as well as primary disease activity and adverse reactions of therapy with glucocorticoid and immunosuppressants up to 24 months.

DETAILED DESCRIPTION:
A total of 120 Chinese patients with connective tissue disease-associated interstitial lung disease (CTD-ILD), including inflammatory myopathy (IIM), rheumatoid arthritis (RA), systemic sclerosis (SSc), and other connective tissue diseases, will be enrolled to use Pirfenidone or not in this study according to 2:1 random entry. Glucocorticoid and immunosuppressants worked as background treatment.

The main research endpoint is the lung function (FVC) at 6 months. The clinical dyspnea score, 6-minute walking distance, lung function and imaging indicators, primary disease activity index are evaluated regularly until 24 months. The relationship of pirfenidone concentration, clinical effect and safety, immune function will be analyzed also.

ELIGIBILITY:
1. Age ≥18 years;
2. Meet several CTD diagnostic criteria (RA, IIM, SSc) and UCTD/IPAF classification criteria;
3. HRCT diagnosis confirmed interstitial lung disease (ILD) with corresponding clinical manifestations;
4. Patients who were able to complete vital capacity (FVC) or carbon monoxide dispersion (DLco) tests (with Hb correction).
5. Patients with clinical deterioration more than 1 month after diagnosis of ILD history, or poor response or intolerance to Glucocorticoids or immunosuppressants treatment, or poor response or intolerance to other antifibrotic drugs (acetyl hemitrine, nidanib, etc.), or effective use of PFD, and exacerbation of clinical symptoms or ILD indicators more than 3 months after withdrawal of the drug.
6. Poor response was defined as no improvement in one of the following:

(1) Symptoms of dyspnea such as cough, chest tightness, breathlessness, shortness of breath after activity, or decreased activity endurance;

(2) the worst decrease in oxygen saturation as measured by pulse oxygen saturation (SpO2) observed during 6MWD;

(3) There was no improvement in pulmonary ventilation (FVC%) or lung dispersion (DLco%);

(4) HRCT findings: new onset, fibrosis tendency or density of ILD lesions were not decreased;

Clinical deterioration was defined as meeting one of three criteria:

1. Clinical deterioration or dyspnea within 4 weeks;
2. New or worsening radiological abnormalities on chest X-ray or high-resolution CT;
3. Objective deterioration of pulmonary function tests or gas exchange, defined as meeting at least one of the following criteria:

1) Start long-term oxygen therapy or increase oxygen supplementation by at least 1 L/min to maintain resting oxygen saturation of at least 90%;

2) FVC decreased by more than 5% compared with the previously measured value; Or a decrease in DLCO of more than 10% from previous measurements; Or a 20% decrease in 6MWD from previous measurements.

7. If concomitant therapy with immunosuppressants was used, the dose was stable for at least 4 weeks before the baseline period. The types of immunomodulator hydroxychloroquine (HCQ) or immunosuppressive agents are MMF, TAC, JAKi, CTX, LEF, AzA, iguratimod etc.

8. Concomitant glucocorticoids: IIM patients with glucocorticoids dose (calculated as the equivalent dose of prednisone) ≤60mg/d and relatively stable disease; For other CTD patients, the glucocorticoids dose (calculated as prednisone equivalent dose) was ≤40mg/ day for at least 1 month.

Exclusion Criteria:

1. Subjects have systemic vasculitis, other arthritis other than CTD or RA such AS psoriatic arthritis, SPA, AS, SLE and pSS;

2. ILD patients with other obvious causes, such as HIV, GVHD, etc.

3. Patients with obvious abnormal combined organ function;

1. Liver :AST, ALT, R-GT, bilirubin at 1.5 ULN, or previously diagnosed viral hepatitis;
2. Kidney: creatinine clearance rate 30ml /min;
3. Lung: airway obstruction (pre-bronchodilator FEV1/FVC & LT; 0.7), pleural effusion accounted for more than 20% of pleural effusion, severe pulmonary infection or other clinically significant pulmonary abnormalities;
4. Cardiovascular: myocardial infarction within 6 months;
5. gastrointestinal tract: active peptic ulcer or bleeding;
6. Blood system: severe anemia, leukopenia, thrombocytopenia;
7. Nervous system: patients with mental disorders; Cerebral thrombotic events (stroke and transient ischemic attack) within the last 1 year;

4. Tuberculosis, cancer, hereditary diseases and other diseases with poor prognosis;

5. Effective contraception cannot be guaranteed during pregnancy, lactation or childbearing age;

6. Evidence of alcohol or drug abuse, according to the researchers;

7. Allergic to glucocorticoids, immunosuppressants and PFD;

8. Unable to complete regular follow-up and post-treatment pulmonary function tests;

9. PFD users not included in the efficacy analysis but included in the safety analysis: those who had used PFD for less than 3 months 6 months before the primary endpoint; The duration of use was less than 3 months before the 24th month of the syudy and the total duration of use was less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in FVC% | 6 months
  change in percentage of forced vital capacity (FVC) from 6 months to baseline

SECONDARY OUTCOMES:
Change in FVC % | 3months 12 months 24 months
  change from baseline in percentage of forced vital capacity (FVC)
change in FEV1%、DLco%、TLC% | 3months 6months 12months 24months
  change from baseline in carbon monoxide diffusing capacity (DLco)、FEV1、TLC
Proportion of patients and time with a decrease in DLco% | 3months 6months 12months 24months
  Percentage of patients and time with DLco% decreased>15% compared to baseline
Proportion of patients and time with a decrease in FVC% | 3months 6months 12months 24months
  Percentage of patients and time with FVC% decreased>10% compared to baseline
Progression-free survival | up to 24months
  survival with a predicated absolute FVC% decrease of no more than 10% from baseline,and a predicated absolute DLco% decrease of no more than 15% from baseline
change in absolute value of FVC and DLco | 3months 6months 12months 24months
  absolute value change of FVC(ml) and DLco(ml) at each time point and annual decline rate compared with baseline
changes from baseline in 6 minutes walking distance | 3months 6months 12months 24months
  changes from baseline in 6 minutes walking distance
change in pulse oxygen saturation | up to 24months
  the worst oxygen saturation as measured by pulse oxygen saturation(SpO2) was observed during 6 minutes walking distance
Worsening respiratory symptoms | 3 months 6months 12months 24months
  Proportion of patients with worsening respiratory symptoms at each time point compared with baseline
Advances in imaging | 3 months 6months 12months 24months
  The proportion of patients with disease progression on imaging at each time point compared with baseline
Imaging changes | 6months 12months 24months
  changes from baseline in high-resolution computed tomography (HRCT)
Borg dyspnea Index score | 3 months 6months 12months 24months
  cChange of Borg dyspnea index score at each time point compared with baseline
clinical deteriorration | up to 24months
  The time and incidence of the first clinical deterioration ,Number of clinical exacerbations,Time between the all-cause deaths
Changes from baseline in C-reactive protein (CRP),Erythrocyte Sedimentation Rate(ESR),Inflammatory factors and indicators. | 3 months 6months 12months 24months
  Changes from baseline in C-reactive protein (CRP),Erythrocyte Sedimentation Rate(ESR),Inflammatory factors and indicators.
Changes from baseline in primary disease activity | up to 24months
  Changes from baseline in primary disease activity
Adverse events , timing,type,extent,frequency,and outcome of SAE | up to 24months
  Adverse events , timing,type,extent,frequency,and outcome of SAE
FVC% area under the curve | 3months 6months 12months 24months
  forced vital capacity (FVC)% area under the curve
Predicators of pirfenidone response in each disease subgroup | 3months 6months 12months 24months
  Predicators of pirfenidone response in each disease subgroup

CONTACTS AND LOCATIONS:
Overall Officials: xiaoyun yang, Dr, Principal Investigator — Study Principal Investigator Qilu HOspital of Shandong Uniwersity
Locations (1):
- Qilu Hospital, Jinan, Shandong, China